CLINICAL TRIAL: NCT06897085
Title: Efficacy of a Gel Containing Polynucleotides and Hyaluronic Acid in the Treatment of Periodontal Supraosseous Defects with the Single Flap Approach: a Randomized Controlled Trial
Brief Title: Efficacy of a Gel Containing Polynucleotides and Hyaluronic Acid in Supraosseous Periodontal Defects Treated with the Single Flap Approach
Acronym: SFA-SD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unità Sanitaria Locale (A.U.S.L.) Ferrara, Italy (Other)
Responsible Party: Principal Investigator, Anna Simonelli, Principal Investigator, Azienda Unità Sanitaria Locale (A.U.S.L.) Ferrara, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7359; Osteology Foundation (Other Grant/Funding Number: Project number: 23-031)
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Gingival Recession, Localized; Aesthetic Perception; Aesthetic Outcomes
Keywords: minimally invasive; single flap approach
MeSH Terms: conditions — Periodontitis; Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Flap Approach (SFA) plus gel containing polynucleotides and hyaluronic acid (PN-HA) (Experimental): Defects treated in this study arm will receive a surgical intervention based on the SFA and will receive the application of PN-HA gel at the completion of defect debridement.
  Interventions: Device: viscoelastic gel containing polynucleotides and hyaluronic acid
- Single Flap Approach (SFA) alone (Sham Comparator): Defects will receive a surgical intervention based on SFA alone (no PN-HA gel will be addedd)
  Interventions: Other: No intervention

INTERVENTIONS:
Device: viscoelastic gel containing polynucleotides and hyaluronic acid — Defects randomized to "test treatment" will receive a viscoelastic gel containing polynucleotides and hyaluronic acid (PN-HA gel) immediately at the completion of intra-surgical instrumentation. PN-HA gel will be also applied on the surgical wound at the completion of the suturing phase.
  Arms: Single Flap Approach (SFA) plus gel containing polynucleotides and hyaluronic acid (PN-HA)
Other: No intervention — Defects randomized to "control group" will be accessed with the SFA and no PN-HA gel will be applied.
  Arms: Single Flap Approach (SFA) alone

SUMMARY:
Treatment of supraosseous defects (SD) may be challenging due to their limited regenerative potential. When located in aesthetic areas, treatment may result in a gingival recession increase with consequent patients' concerns in terms of aesthetic or tooth sensibility. In the present study, a minimally-invasive surgical procedure (namely, the Single Flap Approach, SFA) will be combined with the application of a viscoelastic gel containing polynucleotides and hyaluronic acid that was reported to positively modulate periodontal wound healing. The outcomes, evaluated 6 months after treatment, will be compared to those obtained with SFA alone. The evaluated outcomes will be either clinical (evaluation of clinical parameters such as gingival recession, residual probing depth, clinical attachment gain) or related to patient's perception (such as evaluation of the aesthetic or tooth sensibility).

DETAILED DESCRIPTION:
SDs have been indicated as the most challenging lesions when dealing with periodontal regenerative procedures. In fact, their non-containing morphology does not contribute wound stability, and the wound maturation phase does not benefit from the cellular support coming from residual lateral bony walls, as in intraosseous defects. Also, the absence of residual bony walls does not allow a proper support of the surgical flaps, thus reducing the space needed for regeneration. Because of this unfavorable morphology, treatment of SDs generally results in worse clinical outcomes compared to intraosseous defects. Nevertheless, noteworthy clinical results have been reported when SDs associated to moderate or deep PD were treated with open flap debridement alone. In a systematic review Graziani et al. (2014), showed mean PD reductions of 1.41 mm in sites of moderate pre-surgical pocket depth (i.e., mean PD of 5.19 mm) that reached mean residual pockets of 3.83 mm over 6 months after treatment. More recently, a high prevalence of closed pockets (i.e., 79.3% of sites with residual PD ≤ 3mm) have been reported 12 months after treatment of deep (i.e., mean presurgical value of 6.3 ±0.6 mm) sites with access flap based on papilla preservation techniques (i.e., Modified/Simplified Papilla Preservation Technique).

In 2021, the Single Flap Approach (SFA), a surgical technique originally introduced in the treatment of intraosseous defects, have been also proposed for SDs. The basic principle underlying the SFA is the elevation of a single flap (i.e., on the buccal or oral aspect only, depending on the main extension of the defect) to access the defect, leaving the interproximal supracrestal soft tissue intact. Data stemming from a retrospective analysis showed that the SFA with or without EMD was similarly effective in the treatment deep bleeding pockets associated to a horizontal pattern of bone destruction. In the study arm receiving SFA as a stand-alone protocol, significant mean CAL gains (2.1± 0.9 mm) and PD reductions (3.1± 1.0 mm) were observed 12 months after therapy. These results appear similar or even superior when compared to those reported by other studies where SDs were accessed with Double Flap Approach (based on Papilla Preservation Techniques) alone. Interestingly, this observation has been confirmed by a recent study where clinical and radiographic outcomes observed after surgical access of SDs performed by either a SFA or a DFA were compared. At 6 months, treatment with SFA resulted in greater prevalence of sites reaching CAL gain ≥ 1mm (80% vs 11%) and PD≤ 3mm (40% vs 10%) compared to DFA, thus suggesting that SFA principles may lead to improved clinical outcomes compared to DFA even in the treatment of SDs.

Although the evidence from previous studies support the SFA as a promising treatment for SDs, some clinical aspects currently need further investigation. In the study by Simonelli et al. (2021), a tendency to suboptimal wound closure was evident, with 30% of defects undergoing SFA alone showing Early Healing Index (EHI) scores of 4 or 5 at 2 weeks after surgery. Based on data coming from a previous study demonstrating a trend towards better clinical outcomes (greater CAL gain, less buccal REC increase) in defects with optimal wound closure compared to incomplete wound closure, we may hypothesize that this aspect could have negatively influenced the observed clinical results. In fact, 1-year CAL gain (2.1 mm) was limited if compared to pre-surgery CAL (7.5 mm), and a mean gingival recession (REC) increase of 1 mm was observed.

Recently, a viscoelastic gel containing polynucleotides and hyaluronic acid (PN-HA) was shown to positively influence the viability and proliferation of gingival fibroblasts, thus representing a plausible candidate as periodontal wound modulator. These in vitro results had been partially confirmed by a clinical study where the use of a PN-HA gel showed a higher tendency to pocket closure after subgingival re-instrumentation of PD≥ 5 mm. To date, no clinical data on the effectiveness of PN-HA gel after surgical treatment of SDs is available.

Primary aim The primary aim of the study will be to evaluate the superiority of SFA + PN-HA gel over SFA for the change in interproximal gingival recession (iREC) observed 6 months after surgery of SDs in esthetic areas.

Secondary aims The secondary aims of the study will be to comparatively evaluate SFA + PN-HA gel and SFA for the (i) 6-month prevalence of closed, non-bleeding pockets (i.e., PD≤ 4mm); (ii) quality of early wound closure; (iii) 6-month CAL gain; (iv) 6-month change in buccal gingival recession (bREC); (v) 6-month change in radiographic defect depth; (vi) duration of the surgical procedure; (vii) PROMs, including adverse events, postoperative pain intensity/duration, and patient satisfaction.

ELIGIBILITY:
INCLUSION CRITERIA Patient-specific

* age≥ 18 years;
* diagnosis of Stage III or IV periodontitis22;
* good physical status (ASA1 and ASA2 according to Physical Status Classification System);
* systemic and local conditions compatible with periodontal surgical procedures;
* patient willing and fully capable to comply with the study protocol.

Site-specific

* defect located in an incisor, canine or premolar region which becomes exposed during spontaneous smiling;
* defect with an intrabony component (as assessed on periapical radiograph and confirmed intra-surgically) ≤ 2 mm;
* defect with a radiographic CEJ-BC≥ 4 mm; d) residual (following step I-II of treatment) PD≥6 mm at both interproximal aspects facing the SD.

EXCLUSION CRITERIA Patient-specific

* poorly controlled diabetes (HbA1C ≥ 7%);
* history of radiation therapy in the head and neck area;
* history of chemotherapy;
* systemic disease or conditions with a documented effect on bone metabolism and/or periodontal status/healing;
* past (within 6 months prior to enrollment in the study) or current treatment with any medication with a documented effect on bone metabolism and/or periodontal status/healing;
* physical or mental handicap that can interfere with adherence to the study procedures and adequate hygienic compliance;
* documented allergy to dental materials involved in the experimental protocol;
* pregnancy or lactation;
* history of drug or alcohol abuse.

Moreover, participants will be immediately excluded from the study:

* upon request to withdraw from further participation;
* development of acute dental/periodontal or oral conditions requiring treatment;
* development of conditions conflicting with the exclusion criteria listed above
* failure to comply with study instructions/requirements.

Site-specific

* presence of untreated endodontic lesions or inadequate endodontic treatment of teeth facing the SD;
* presence of orthodontic appliances;
* local conditions preventing proper plaque control at experimental sites;
* grade III mobility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Interproximal gingival recession (iREC) | 6 months after surgical treatment of supraosseous defects
  the primary outcome of the study will be iREC change

SECONDARY OUTCOMES:
Prevalence of closed, non bleeding pockets | 6 months after surgical treatment
  closed pocket (i.e., residual 6-month probing depth (PD)≤ 4mm)
Quality of early wound closure | 2-week follow-up
  The quality of early wound closure will be evaluated using the "early healing index" (EHI), as proposed by Wachtel et al. in 2003.
  EHI is based on the following scale: (EHI=1) complete flap closure, no fibrin line in the interproximal area; (EHI=2) complete flap closure, fine fibrin line in the interproximal area; (EHI=3) complete flap closure, fibrin clot in the interproximal area; (EHI=4) incomplete flap closure, partial necrosis of the interproximal tissue; and (EHI=5) incomplete flap closure, complete necrosis of the interproximal tissue.
Clinical Attachment Level (CAL) Gain | 6 months after surgical treatment
  6-month CAL gain will be calculated by subtracting the 6-month CAL value from the baseline CAL
Change in buccal gingival recession (bREC); | 6 months after surgical treatment
  bREC change will be calculated by subtracting the 6-month bREC value from the baseline bREC value
Change in radiographic defect depth | 6 months after surgical treatment
  change in radiographic defect depth will be calculated by subtracting the 6-month radiographic defect depth value from the baseline radiographic defect depth value
PROMs | post-operative days 1, 2, 7 and 14
  PROMs will include adverse events, postoperative pain intensity/duration, and patient satisfaction.
  Both "postoperative course" and "patient satisfaction" will be assessed through a self-administered questionnaire and/or a VAS (1-100) ranging from "0 - no pain/no satisfaction" to "100 - intolerable pain/full satisfaction".

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graziani F, Gennai S, Cei S, Ducci F, Discepoli N, Carmignani A, Tonetti M. Does enamel matrix derivative application provide additional clinical benefits in residual periodontal pockets associated with suprabony defects? A systematic review and meta-analysis of randomized clinical trials. J Clin Periodontol. 2014 Apr;41(4):377-86. doi: 10.1111/jcpe.12218. Epub 2014 Jan 22. PMID 24329867
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Papapanou PN, Wennstrom JL. The angular bony defect as indicator of further alveolar bone loss. J Clin Periodontol. 1991 May;18(5):317-22. doi: 10.1111/j.1600-051x.1991.tb00435.x. PMID 2066446
- [Background] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787
- [Background] Simonelli A, Minenna L, Trombelli L, Farina R. Single flap approach with or without enamel matrix derivative in the treatment of severe supraosseous defects: a retrospective study. Clin Oral Investig. 2021 Nov;25(11):6385-6392. doi: 10.1007/s00784-021-03941-5. Epub 2021 Apr 14. PMID 33855656
- [Background] Trombelli L, Farina R, Franceschetti G, Calura G. Single-flap approach with buccal access in periodontal reconstructive procedures. J Periodontol. 2009 Feb;80(2):353-60. doi: 10.1902/jop.2009.080420. PMID 19186978